CLINICAL TRIAL: NCT07190391
Title: A Multi-center, Single-arm, Open-label, Phase 4 Clinical Study to Evaluate the Efficacy and Safety of Apremilast in Patients With Moderate-to-severe Psoriasis
Brief Title: Phase 4 Multicenter, Open-label Study on Efficacy and Safety of Apremilast in Moderate-to-severe Psoriasis
Status: Not yet recruiting | Type: Observational
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: DWAPS_P401
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Apsola Tab.: Apsola Tab. 10mg, Apsola Tab. 20mg, Apsola Tab. 30mg

SUMMARY:
This study aims to evaluate the efficacy and safety of Apremilast tablets in patients with psoriasis over 32 weeks, through a multicenter, single-arm, open-label, phase 4 clinical trial.

DETAILED DESCRIPTION:
In this clinical trial, patients with psoriasis will be informed about study participation and written informed consent will be obtained voluntarily. Eligible participants, based on inclusion and exclusion criteria, will be assigned a registration number. Participants will receive Apremilast for 32 weeks and visit the study site at three time points: Visit 1 (screening and baseline, Week 0), Visit 2 (Week 16 ± 4), and Visit 3 (Week 32 ± 4). At each visit, demographic information, efficacy assessments, and adverse event evaluations will be conducted according to the study schedule.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥19 years at the time of enrollment.
* Patients with moderate to severe psoriasis persisting for ≥6 months.
* Patients with a PASI (Psoriasis Area and Severity Index) score between 5 and 10, requiring pharmacological treatment.
* Patients who have been fully informed about the study, have understood the explanation, and have voluntarily signed the informed consent form.
* Patients who are considered cooperative and able to participate until the end of the study.

Exclusion Criteria:

* Patients with a history of hypersensitivity to apremilast.
* Patients with genetic disorders such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
* Pregnant or breastfeeding women.
* Patients (or their spouse/partner) who do not agree to use medically acceptable and appropriate methods of contraception* during the study period.

  * Medically acceptable and appropriate methods of contraception include: hormonal contraception (implants, injectables, oral contraceptives, etc.), intrauterine devices (copper IUD, hormone-releasing intrauterine system), salpingectomy, tubal ligation, hysterectomy, vasectomy, dual barrier methods (male condom and female condom, cervical cap, diaphragm, contraceptive sponge used in combination), or single barrier method combined with spermicide.
* Patients receiving strong CYP3A4 enzyme inducers (e.g., rifampicin, phenobarbital, carbamazepine, phenytoin, St. John's Wort).
* Patients with severe renal impairment requiring hemodialysis or peritoneal dialysis.
* Patients who have previously received Apremilast (ApsoLla®) prior to enrollment, or those currently participating in another clinical trial involving an investigational medicinal product or medical device.

(However, patients enrolled in non-interventional studies or who have completed participation in another clinical trial are eligible.)

* Patients with a history of psychiatric disorders (e.g., substance abuse, depression).
* Patients who, in the opinion of the investigator, are otherwise considered unsuitable for participation in this study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the ESTEEM 1 study of moderate-to-severe psoriasis, 33.1% of patients achieved PASI 75 at Week 16 with apremilast, while 28.8% did so in ESTEEM 2. Based on these results, this trial assumed a Week 16 PASI 75 response rate of ~30%. To estimate this with a 95% confidence interval and ±5% margin of error, a sample size of 340 was calculated. If the observed rate is 30%, the Clopper-Pearson method yields a lower bound of 25.2%. The study aims to present the Week 16 PASI 75 response rate with 95% confidence in a single-arm design, ensuring effect size and precision. Considering ~20% dropout, 425 subjects will be enrolled.
Sampling Method: Probability Sample
Enrollment: 425 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who achieved PASI 75 | 16 weeks
  Proportion of patients who achieved PASI 75 at week 16

SECONDARY OUTCOMES:
[Investigator-Assessed Endpoints]Proportion of patients who achieved PASI 75 | 32 weeks
  Proportion of patients who achieved PASI 75 at week 32
[Investigator-Assessed Endpoints]Proportion of patients who achieved PASI 50 | 16 weeks
  Proportion of patients who achieved PASI 50 at weeks 16
[Investigator-Assessed Endpoints]Proportion of patients who achieved PASI 50 | 32 weeks
  Proportion of patients who achieved PASI 50 at weeks 32
[Investigator-Assessed Endpoints]Proportion of patients who achieved PASI 90 | 16 weeks
  Proportion of patients who achieved PASI 90 at weeks 16
[Investigator-Assessed Endpoints]Proportion of patients who achieved PASI 90 | 32 weeks
  Proportion of patients who achieved PASI 90 at weeks 32
[Investigator-Assessed Endpoints]Proportion of patients with an absolute PASI score ≤ 2 | 16 weeks
  Proportion of patients with an absolute PASI score ≤ 2 at weeks 16
[Investigator-Assessed Endpoints]Proportion of patients with an absolute PASI score ≤ 2 | 32 weeks
  Proportion of patients with an absolute PASI score ≤ 2 at weeks 32
[Investigator-Assessed Endpoints]Percentage improvement in mNAPSI (modified Nail Psoriasis Severity Index) | 16 weeks
  Percentage improvement in mNAPSI (modified Nail Psoriasis Severity Index) from baseline at weeks 16
[Investigator-Assessed Endpoints]Percentage improvement in mNAPSI (modified Nail Psoriasis Severity Index) | 32 weeks
  Percentage improvement in mNAPSI (modified Nail Psoriasis Severity Index) from baseline at weeks 32
[Investigator-Assessed Endpoints]Proportion of patients who achieved ScPGA (Scalp Physician Global Assessment) score of 0 or 1 | 16 weeks
  Proportion of patients who achieved ScPGA (Scalp Physician Global Assessment) score of 0 or 1 at weeks 16
[Investigator-Assessed Endpoints]Proportion of patients who achieved ScPGA (Scalp Physician Global Assessment) score of 0 or 1 | 32 weeks
  Proportion of patients who achieved ScPGA (Scalp Physician Global Assessment) score of 0 or 1 at weeks 32
[Patient-Reported Endpoints]Change from baseline in DLQI (Dermatology Life Quality Index) | 16 weeks
  Change from baseline in DLQI (Dermatology Life Quality Index) at weeks 16
[Patient-Reported Endpoints]Change from baseline in DLQI (Dermatology Life Quality Index) | 32 weeks
  Change from baseline in DLQI (Dermatology Life Quality Index) at weeks 32
[Patient-Reported Endpoints]Change from baseline in Pruritus NRS (Numeric Rating Scale) | 16 weeks
  Change from baseline in Pruritus NRS (Numeric Rating Scale) at weeks 16
Change from baseline in Pruritus NRS (Numeric Rating Scale) | 32 weeks
  Change from baseline in Pruritus NRS (Numeric Rating Scale) at weeks 32
[Patient-Reported Endpoints]Change from baseline in PaGA (Patient Global Assessment) | 16 weeks
  Change from baseline in PaGA (Patient Global Assessment) at weeks 16
[Patient-Reported Endpoints]Change from baseline in PaGA (Patient Global Assessment) | 32 weeks
  Change from baseline in PaGA (Patient Global Assessment) at weeks 32
[Patient-Reported Endpoints]Shift in distribution of PaGA scores | 16 weeks
  Shift in distribution of PaGA scores from baseline at weeks 16
[Patient-Reported Endpoints]Shift in distribution of PaGA scores | 32 weeks
  Shift in distribution of PaGA scores from baseline at weeks 32
[Patient-Reported Endpoints]Proportion of patients who achieved PaGA score of 0 or 1 | 16 weeks
  Proportion of patients who achieved PaGA score of 0 or 1 at weeks 16
[Patient-Reported Endpoints]Proportion of patients who achieved PaGA score of 0 or 1 | 32 weeks
  Proportion of patients who achieved PaGA score of 0 or 1 at weeks 32